CLINICAL TRIAL: NCT03376711
Title: Development & Pilot Randomized Control Trial (RCT) of an Online Peer Support Program for Family Caregivers of Ventilator-Assisted Individuals Living in the Community
Brief Title: Development & Pilot RCT of an Online Peer Support Program for Family Caregivers of Ventilator-Assisted Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Louise Rose, Associate Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 32210
Record Dates: First submitted 2017-05-02; First posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Social Support; Affect; Ventilators, Mechanical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care Group (No Intervention): Participants in this arm of the study will not have access to the online peer support program until the end of the 12-week trial.
- Online Peer Support Program (Experimental): Participants in the online peer support program arm of the intervention will have access to the website for 12 weeks.
  Interventions: Behavioral: Online Peer Support Program

INTERVENTIONS:
Behavioral: Online Peer Support Program — The online peer support program will entail: 1) Informational links; 2) A discussion forum (open to all participants and allowing for asynchronous contact between caregivers & peer mentors); 3) A weekly live chat; 4) Private messaging (audio, video, and text options); and 5) "Ask-a-mentor" (A short video/blurb profiling each caregiving mentor will be posted including details such as gender, age, duration of care, relationship to care-recipient, and illness that care-recipient suffers from). Caregiving participants can then self-match to a peer mentor they feel is best-positioned to address their support needs.
  Arms: Online Peer Support Program

SUMMARY:
Ventilator assisted individuals (VAIs) living at home are frail and generally cannot perform most daily activities. Although these individuals prefer to live at home, the family members who care for them often experience stress and poor health. Peer support can mitigate health declines by decreasing caregivers' isolation/stress and increasing their sense of control. However, no peer support programs are designed to meet these caregivers' complex and unique needs. Online support delivery is especially beneficial for caregivers given the geographic and time limitations they face. The proposed research aims to develop and conduct an RCT of online peer support program for VAI caregivers. A group of caregivers will be trained to act as peer mentors. This training program will be evaluated for its impact on caregivers' mentoring abilities. At the end of the 12-week program, caregiving participants will be asked about the online delivery of the program, how helpful/satisfactory it was, and if it affected their health and well-being. The health outcomes of the control and intervention group will be compared. This peer support program can improve the well-being of caregivers and allow them to better care for their family members.

ELIGIBILITY:
Inclusion Criteria:

1) age = 18 years; 2) primary family caregiver for a VAI living in the community; 3) able to speak and read English; and 4) access to a computer and a reliable internet connection.

Exclusion Criteria:

1) currently experiencing severe depression as indicated by a score of 40 or higher on the Centre for epidemiological studies short depression scale (CES-D 10).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Change in Positive and Negative Affect | Change from baseline at 12 weeks
  Positive & Negative Affect Scale (PANAS): 10 items [Score: 10-50]; higher scores indicate more psychological wellbeing

SECONDARY OUTCOMES:
Feasibility: Participation rate | 12 weeks
  Proportion of mentors and caregiving participants who contribute to weekly chats and discussion forums for all 12 weeks of the program
Feasibility: Participation frequency | 12 weeks
  Number of times that mentors and caregiving participants contribute to weekly chat and discussion forums over the course of 12 weeks. ).
Feasibility: Recruitment rates | Through study completion, an average of 1 year
  Consent rate for participation (i.e. proportion of individuals approached who consent to participate)
Feasibility: Attrition | 12 weeks
  Attrition rates (i.e. number of mentors and caregiving participants who participate in entire peer support program and complete required study questionnaires).
Change in Coping | Change from baseline at 12 weeks
  Brief Coping Orientations to Problems Experienced (COPE) Inventory: 28 items representing problem and emotion-based coping. Higher scores on either subscale represent greater use of that coping style
Change in Depression | Change from baseline at 12 weeks
  ) Centre for Epidemiological Studies Short Depression Scale (CES-D 10): 10 items [Score: 0-30]; higher scores sores indicate depression severity
Change in Caregiving Impact | Change from baseline at 12 weeks
  Caregiving Impact Scale: 14 items [Score: 0-84]; higher scores suggest providing care interferes with caregivers' abilities to maintain participation in valued activities
Change in Mastery | Change from baseline at 12 weeks
  Pearlin Mastery Scale: 7 items [Score: 7-28]; higher scores indicate a greater sense of control over life
Change in Personal Gain | Change from baseline at 12 weeks
  Personal Gain Scale: 4 items [Score: 4-16]; higher scores indicate caregiver discovery of inner strengths due to providing care

CONTACTS AND LOCATIONS:
Overall Officials: Marina B Wasilewski, PhD, Principal Investigator — University of Toronto; Louise Rose, PhD, Principal Investigator — University of Toronto
Locations (1):
- Ventilator Equipment Pool (Queens University), Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No